CLINICAL TRIAL: NCT00118001
Title: Worry Exposure Versus Applied Relaxation in the Treatment of Generalized Anxiety Disorder
Brief Title: Psychotherapy of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HO 1900/3-1, HO 1900/3-2
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2005-06

CONDITIONS: Anxiety Disorders
Keywords: Psychotherapy; Generalized Anxiety Disorder; randomized-controlled trial; worry exposure; applied relaxation
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

INTERVENTIONS:
Behavioral: Worry exposure
Behavioral: Applied relaxation

SUMMARY:
The purpose of this study is to compare the effects of worry exposure with the effects of applied relaxation in patients with generalized anxiety disorder.

DETAILED DESCRIPTION:
Controlled treatment studies show that there is a lower efficacy of cognitive-behavioral treatment of generalized anxiety disorder (GAD) than in other anxiety disorders. The best effect sizes are found for applied relaxation (Öst), but there are only three treatment studies. Another, yet previously not tested in its pure form, approach is "worry-exposure", which aims at confronting the emotionally intensive imaginative contents of worries in GAD.

Fifty-two randomized patients with GAD as a primary diagnosis will be treated with one of the two treatments and will be compared with waiting-list patients. This treatment protocol contains 15 sessions (+/-2) and a 6 month and 12 month follow-up.

The comparisons in this study include: worry exposure versus applied relaxation versus a waiting control group.

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of generalized anxiety disorder (according to impairment)
* 18-70 years of age
* Informed consent

Exclusion Criteria:

* Not able to understand and speak the German language
* Acute, unstable and severe somatic disease (DSM-IV, Axis III)
* History of schizophrenia or bipolar disorder
* Other mental disorders requiring treatment
* Substance dependence within the past 12 months preceding treatment
* Personality disorders that interfere with treatment compliance
* Participation in any other psychotherapeutic interventions
* Use of anxiolytics (e.g. tranquilizer, hypnotics, neuroleptics; does not include stabile use of antidepressants)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2001-10; Study Completion 2006-07

PRIMARY OUTCOMES:
At post-treatment: anxiety (Hamilton Anxiety Rating Scale, HARS), depression (Hamilton Depression Scale, HAM-D), trait-anxiety (State-Trait-Anxiety Inventory, STAI-T)
At 6-month follow-up: M-CIDI (Composite International Diagnostic Interview, generalized anxiety disorder section)

SECONDARY OUTCOMES:
At post-treatment, 6 and 12 month follow-ups:
worry (Penn State Worry Questionnaire, PSWQ)
general symptoms (Brief Symptom Inventory, BSI)
depression (Beck Depression Inventory, BDI)
interpersonal problems (Inventory of Interpersonal Problems - IIP)
meta-cognitions (Meta Cognitions Questionnaire)
thought suppression (White Bear Suppression Inventory) tolerance for uncertainty (Ungewissheitstoleranzskala, UGTS)
positive and negative affect (Positive and Negative Affect Schedule, PANAS)
At post-treatment: behavior assessment tests

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Hoyer, PhD, Principal Investigator — Technische Universität Dresden; Eni S Becker, PhD, Principal Investigator — University of Nijmegen
Locations (1):
- Technische Universität Dresden, Dresden, Germany